CLINICAL TRIAL: NCT00807495
Title: A Phase 2 Trial of MLN8237, an Oral Aurora A Kinase Inhibitor, in Adult Patients With Aggressive Non-Hodgkin's Lymphoma
Brief Title: Study of Alisertib (MLN8237) in Adults With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14004; U1111-1187-1268 (Registry Identifier: WHO)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma; Burkitt's Lymphoma; T-cell Lymphoma, Excluding Primary Cutaneous T-cell Lymphoma; Transformed Follicular Lymphoma With ≥ 50% Diffuse Large Cell Component
Keywords: MLN8237; Alisertib; Drug therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, T-Cell | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib 50 mg (Experimental): Alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 24 months or longer with Sponsor approval).
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib capsules
  Other Names: MLN8237

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity of alisertib (MLN8237) in participants with relapsed or refractory non-hodgkin's lymphoma.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat people who have relapsed or refractory non-Hodgkin's lymphoma (NHL). The study looked at anti-tumor activity in participants who received alisertib.

The study enrolled 48 patients. Participants were categorized as per disease subtypes into five subtypes: Large B-Cell lymphoma, mantle cell lymphoma, transformed follicular lymphoma, Burkitts lymphoma and aggressive T-Cell lymphoma (Note: There were no participants enrolled with Precursor B-lymphoblastic Leukemia/Lymphoma). Participants received:

• Alisertib 50 mg BID on Days 1 to 7

All participants took alisertib capsules approximately every 12 hours each day for 7 days followed by a 14-day rest period in a 21-days cycle. MLN8237 was supplied in capsules of 5 or 25 mg strength.

This multi-center trial was conducted in United States. The overall time to participate in this study was until there is evidence of disease progression or unacceptable treatment-related toxicity. If the participant would derive benefit from continued alisertib treatment beyond 24 months, the Sponsor was consulted for approval of further treatment. Participants made multiple visits to the clinic, with imaging assessments every 12 weeks. Participants discontinuing treatment prior to disease progression continue with clinic visits, chemistry and hematology lab testing, and tumor assessments every 12 weeks up to 12 months after last dose of study drug for follow-up assessments.

ELIGIBILITY:
Each participant must meet all of the following inclusion criteria to be enrolled in the study:

1. Participant must have histological or cytological diagnosis of a hematological malignancy of the following types that has relapsed or was refractory to prior therapy:

   * Diffuse large B-cell lymphoma
   * Mantle cell lymphoma
   * Burkitt's lymphoma
   * Precursor B-lymphoblastic leukemia/lymphoma
   * T-cell lymphoma, excluding primary cutaneous T-cell lymphoma
   * Transformed follicular lymphoma with ≥ 50% diffuse large cell component.
2. Male or female participants 18 years or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Measurable disease.

Exclusion criteria include the following:

1. Pregnant or lactating females.
2. Known human immunodeficiency virus (HIV) positive or AIDS-related illness.
3. Any serious medical or psychiatric illness that could interfere with the completion of treatment.
4. Total bilirubin ≥ 1.5 × the upper limit of normal (ULN).
5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 2.5 × the ULN. AST, ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to their underlying hematological disorder.
6. Absolute neutrophil count (ANC) < 1,250/mm^3.
7. Platelet count < 75,000/mm^3.
8. Calculated creatinine clearance < 30 mL/minute.
9. Autologous stem cell transplant less than 6 months prior to enrollment.
10. Participants who have undergone allogeneic stem cell or organ transplantation.
11. Systemic antineoplastic therapy including glucocorticoids (> 15 mg prednisone/day or equivalent), or treatment with an investigational agent within 14 days preceding the first dose of study drug treatment.
12. Participants who have received treatment with nitrosoureas, mitomycin C, rituximab, alemtuzumab, or other unconjugated antibody treatment, within 12 weeks prior to first dose.
13. Participants who have received treatment with radioimmunoconjugates or within 12 weeks prior to first dose.
14. Participants who have received radiotherapy within 21 days prior to first dose.
15. Myocardial infarction within 6 months of enrollment or current history of New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
16. Major surgery within 14 days prior to the first dose.
17. Infection requiring systemic antibiotic therapy within 14 days prior to the first dose or other serious infection.
18. Clinically uncontrolled central nervous system (CNS) involvement.
19. Inability to swallow capsules.
20. History of uncontrolled sleep apnoea syndrome and other conditions that could result in excessive daytime sleepiness (eg, Chronic obstructive pulmonary disease - COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02-10 (Actual); Primary Completion 2011-01-04 (Actual); Study Completion 2013-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Hematology Oncology Associates, Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey, United States

REFERENCES:
- [Result] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in the United States from 10 February 2009 to last participant off study 13 February 2013, with a data cut-off on 04 January 2011 to report the primary endpoint.
Pre-assignment Details: Participants with a diagnosis of Aggressive Non-Hodgkin's Lymphoma received 50 mg alisertib twice daily for 7 days in 21 day cycles. Results are categorized as disease sub-types: Diffuse Large B-cell lymphoma (DLBL), Mantle Cell lymphoma (MCL), Transformed Follicular lymphoma (TFL), Burkitts lymphoma (BL) and Aggressive T-Cell lymphoma (ATL).
Groups:
- Alisertib 50 mg BID Starting Dose (DLBL): Participants with diffuse large B-Cell lymphoma (DLBL) received alisertib 50 mg, capsules, orally, twice daily (BID) for 7 days, followed by 14-day rest period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 24 months).
- Alisertib 50 mg BID Starting Dose (MCL): Participants with mantle cell lymphoma (MCL) received alisertib 50 mg, capsules, orally, BID for 7 days, followed by 14-day rest period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 24 months).
- Alisertib 50 mg BID Starting Dose (TFL): Participants with transformed follicular lymphoma (TFL) received alisertib 50 mg, capsules, orally, BID for 7 days, followed by 14-day rest period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 24 months).
- Alisertib 50 mg BID Starting Dose (BL): Participants with Burkitts lymphoma (BL) received alisertib 50 mg, capsules, orally, BID for 7 days, followed by 14-day rest period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 24 months).
- Alisertib 50 mg BID Starting Dose (ATL): Participants with aggressive T-Cell lymphoma (ATL) received alisertib 50 mg, capsules, orally, BID for 7 days, followed by 14-day rest period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 24 months).
Period: Overall Study
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Started | 22 | 13 | 5 | 1 | 7 (An ATL participant had late on-study biopsy and was in DLBL, reducing ATL participants from 8 to 7.)
Completed | 14 (Completed = participants who completed the study treatment to PD or symptomatic deterioration.) | 7 | 1 | 0 | 2
Not Completed | 8 | 6 | 4 | 1 | 5
Not completed — Adverse Event | 6 | 3 | 1 | 1 | 2
Not completed — Withdrawal by Patient | 2 | 0 | 1 | 0 | 0
Not completed — Reason Not Specified | 0 | 3 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received any amount of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL) | Total
Number analyzed (Participants) | 22 | 13 | 5 | 1 | 7 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (11.11) | 67.2 (6.71) | 65.2 (9.96) | 76.0 (NA) — Standard deviation was not estimable as only 1 participant was analyzed in this arm group. | 54.4 (16.90) | 65.1 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 3 | 0 | 0 | 13
  Male | 13 | 12 | 2 | 1 | 7 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 13 | 5 | 1 | 7 | 47
  Other | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 21 | 13 | 4 | 1 | 6 | 45
Weight [Mean (Standard Deviation); unit: kg] | 88.85 (27.022) | 96.18 (25.139) | 89.06 (29.724) | 72.58 (NA) — Standard deviation was not estimable as only 1 participant was analyzed in this arm group. | 84.45 (14.494) | 89.88 (24.737)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate Based on Investigator's Assessment (Applying the IWG 2007 Response Criteria)
Description: Best overall response rate is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the Investigator using International Working Group (IWG) Criteria. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites (as specified in the Cheson 2007, IWG response criteria).
Time Frame: Baseline and every 2 cycles up to Month 12 (approximately 16 cycles), from Cycle 16 every 4 cycles until disease progression, after end of treatment every 12 weeks for up to 12 Months from last dose (Up to 4 years)
Population: Safety population was defined as all participants who received any amount of alisertib. Efficacy analysis for the response-evaluable population is a subset of the safety population, with participants having a minimum of baseline imaging and one on-study imaging.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 16 | 13 | 5 | 1 | 6
percentage of participants | 25 | 23 | 40 | 100 | 50

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) is defined as the time in days from the date of first study drug administration to the date of first documentation of Progressive Disease (PD) according to IWG criteria (Cheson 2007). PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: Baseline and every 2 cycles up to Month 12, from Cycle 16 every 4 cycles until disease progression, after end of treatment every 12 weeks for up to 12 Months (Up to 4 years)
Population: Response-evaluable population is subset of safety population, defined as all participants who received any amount of alisertib, having minimum of baseline imaging and one on-study imaging. Here number of participants analyzed were participants with PD. TTP was censored at the last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 16 | 13 | 5 | 1 | 6
days | 84.0 [48.0 to 430.0] | 139.0 [48.0 to 809.0] | NA [NA to NA] — Median was not reached due to the low number of participants with events. | NA [NA to NA] — Median was not reached due to the low number of participants with events. | 237.0 [46.0 to 631.0]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in days from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death.
Time Frame: as for outcome 2
Population: Response-evaluable population is subset of safety population, defined as all participants who received any amount of alisertib, having minimum of baseline imaging and one on-study imaging. For a participant who had not progressed and had not died, PFS was censored at the last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 16 | 13 | 5 | 1 | 6
days | 84.0 [48.0 to 364.0] | 139.0 [48.0 to 809.0] | NA [NA to NA] — Median was not reached due to the low number of participants with events. | NA [NA to NA] — Median was not reached due to the low number of participants with events. | 237.0 [46.0 to 631.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a CR, or partial response (PR) to the date of first documentation of PD according to IWG criteria. CR definition includes the complete disappearance of all evidence of disease, the definition of PR includes at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses, and PD is defined as any new lesion or increase by >50% of previously involved sites from nadir, as described in the IWG response criteria (Cheson 2007).
Time Frame: as for outcome 2
Population: Response-evaluable population is subset of safety population, defined as all participants who received any amount of alisertib, having minimum of baseline imaging and one on-study imaging. All responders were evaluated in this outcome measure. Participants who had not progressed, DOR was censored at last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 4 | 3 | 2 | 1 | 3
days | 454.0 [182.0 to 565.0] | 646.0 [243.0 to 646.0] | NA [NA to NA] — Median was not reached due to the low number of participants with events. | NA [NA to NA] — Median was not reached due to the low number of participants with events. | 596.0 [202.0 to 596.0]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug and includes all-causality (ie, treatment-related and not treatment-related as assessed by the investigator).
Time Frame: First dose of study drug to 30 days after last dose (Up to 25 months)
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 22 | 13 | 5 | 1 | 7
participants | 22 | 13 | 5 | 1 | 7

6. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events
Description: Vital signs (blood pressure, heart rate, and oral temperature) measurements were obtained throughout the study. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after last dose (Up to 25 months)
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 22 | 13 | 5 | 1 | 7
participants
  Pyrexia | 7 | 0 | 0 | 0 | 2
  Hypotension | 6 | 1 | 1 | 0 | 1
  Weight decreased | 2 | 1 | 0 | 0 | 1
  Tachycardia | 1 | 0 | 0 | 0 | 2
  Hypertension | 1 | 0 | 0 | 0 | 0
  Bradycardia | 1 | 0 | 0 | 0 | 0
  Cardiac flutter | 1 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Laboratory Values Reported as Treatment-Emergent Adverse Events
Description: Abnormal laboratory values for chemistry or hematology tests that were assessed by the investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE V4). A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after last dose (Up to 25 months)
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Number analyzed (Participants) | 22 | 13 | 5 | 1 | 7
participants
  Thrombocytopenia | 11 | 5 | 3 | 1 | 5
  Alanine aminotransferase increased | 6 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 6 | 0 | 0 | 0 | 1
  Blood alkaline phosphatase increased | 6 | 0 | 0 | 0 | 1
  Hypokalaemia | 3 | 0 | 1 | 0 | 1
  Blood lactate dehydrogenase increased | 3 | 0 | 0 | 0 | 1
  Blood creatinine increased | 0 | 0 | 0 | 0 | 2
  Blood potassium decreased | 1 | 0 | 0 | 0 | 1
  Lymphopenia | 1 | 0 | 0 | 0 | 1
  Blood urea increased | 1 | 0 | 0 | 0 | 0
  Hypercalcaemia | 0 | 0 | 0 | 0 | 1
  Hypernatraemia | 0 | 0 | 0 | 0 | 1
  Hypophosphataemia | 0 | 0 | 0 | 0 | 1
  Mean cell volume increased | 0 | 0 | 0 | 0 | 1
  Urine colour abnormal | 0 | 1 | 0 | 0 | 0
  Neutropenia | 13 | 9 | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose (Up to 25 Months)
Description: The investigator documents any occurrence of adverse events including abnormal laboratory findings. Additionally, any event spontaneously reported by the participant or observed by the investigator are recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib 50 mg BID Starting Dose (DLBL) | Alisertib 50 mg BID Starting Dose (MCL) | Alisertib 50 mg BID Starting Dose (TFL) | Alisertib 50 mg BID Starting Dose (BL) | Alisertib 50 mg BID Starting Dose (ATL)
Serious Adverse Events (participants affected / at risk) | 16/22 | 4/13 | 5/5 | 0/1 | 4/7
Other Adverse Events (participants affected / at risk) | 22/22 | 13/13 | 5/5 | 1/1 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg BID Starting Dose (DLBL) (N=22) | Alisertib 50 mg BID Starting Dose (MCL) (N=13) | Alisertib 50 mg BID Starting Dose (TFL) (N=5) | Alisertib 50 mg BID Starting Dose (BL) (N=1) | Alisertib 50 mg BID Starting Dose (ATL) (N=7)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg BID Starting Dose (DLBL) (N=22) | Alisertib 50 mg BID Starting Dose (MCL) (N=13) | Alisertib 50 mg BID Starting Dose (TFL) (N=5) | Alisertib 50 mg BID Starting Dose (BL) (N=1) | Alisertib 50 mg BID Starting Dose (ATL) (N=7)
Neutropenia (Blood and lymphatic system disorders) | 16 | 9 | 4 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 15 | 7 | 3 | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 13 | 8 | 3 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 5 | 3 | 1 | 5
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 8 | 3 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 7 | 2 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 6 | 2 | 1 | 0 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3 | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 12 | 9 | 4 | 0 | 6
Asthenia (General disorders) | 5 | 1 | 2 | 0 | 3
Oedema peripheral (General disorders) | 4 | 1 | 1 | 0 | 2
Pyrexia (General disorders) | 6 | 0 | 0 | 0 | 2
Catheter site erythema (General disorders) | 3 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 8 | 4 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 9 | 4 | 2 | 1 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 6 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 0 | 0 | 0 | 3
White blood cell count decreased (Investigations) | 3 | 1 | 0 | 0 | 2
Haemoglobin decreased (Investigations) | 4 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio decreased (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urine colour abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 2 | 0 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 3 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2
Attention deficit (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 6 | 1 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0
Night blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 2 | 3 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.